CLINICAL TRIAL: NCT06566196
Title: Invasive Hemodynamic Cardiopulmonary Exercise Testing for Assessment of Patients With Congenital Heart Disease (Cath CHD)
Brief Title: A Study of Hemodynamic Cardiopulmonary Exercise for CHD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Alexander C. Egbe, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 24-004619; 5R01HL160761-03 (NIH)
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients Undergoing Clinically indicated Cardiac Cath (Experimental)
  Interventions: Procedure: Cardiac Cath

INTERVENTIONS:
Procedure: Cardiac Cath — Patient will undergo standard of care Cardiac Cath and in addition invasive CPET (Cardiopulmonary exercise testing) will be performed during the procedure.

SUMMARY:
The purpose of this study is to compare the difference in the ability to detect hemodynamic abnormalities between invasive hemodynamic assessments performed at rest versus exercise, to assess the correlation between invasive and noninvasive (Doppler-derived) rest-exercise hemodynamic indices and to compare the association between indices of disease severity and hemodynamic abnormalities identified at rest versus exercise.

ELIGIBILITY:
Inclusion Criteria:

* Congenital Heart Disease Diagnosis
* Undergoing Clinically indicated Cardiac Cath

Exclusion Criteria:

* Unable to consent
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in left ventricular end-systolic elastance from rest to peak exercise | Baseline
  Change in left ventricular end-systolic elastance will be measured in ΔmmHg/mL
Change in Left ventricular cardiac output from rest to peak exercise | Baseline
  Change in left ventricular cardiac output will be measured in ΔL/min
Change in systemic vascular resistance from rest to peak exercise | Baseline
  Change in systemic vascular resistance will be measured in ΔWoods Units
Change in right ventricular free-wall strain from rest to peak exercise | Baseline
  Change in right ventricular free-wall strain will be measured in Δ%
Change in right ventricular cardiac output from rest to peak exercise | Baseline
  Change in right ventricular cardiac output will be measured in ΔL/min
Change in pulmonary vascular resistance from rest to peak exercise | Baseline
  Change in pulmonary vascular resistance will be measured in ΔWoods Units

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Egbe, M.B.B.S., M.P.H., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No